CLINICAL TRIAL: NCT05570604
Title: Computerized Cognitive Training in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Indiana University (Other)
Responsible Party: Principal Investigator, Diane Von Ah, Distinguished Professor of Cancer Research, College of Nursing Director of Cancer Research Center for Healthy Aging, Self-Management and Complex Care, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUSCC-0625
Record Dates: First submitted 2021-12-15; First posted 2022-10-06 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Cognitive Change; Cognitive Impairment; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The purpose of this translational research is to conduct a home based single-blind, randomized controlled trial to test the feasibility, satisfaction, and preliminary efficacy of cognitive training compared to attention control in breast cancer survivors (BCS) as well as to explore potential biomarkers of intervention effects.
Who Masked: Care Provider
Masking Description: A blinded and trained tester will perform data collection and neuropsychological testing at two time points
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): As tested in the investigator's pilot, the Brain HQ program is designed to enhance specific areas of cognitive functioning that will be tested in this study. The goals of the Brain HQ program are to improve visual processing speed, learning and memory and attention. The exercises include time-order judgment, discrimination, spatial-match, forward-span, instruction-following, and narrative-memory tasks. This program systematically reduces the stimulus duration during a series of increasingly difficult information-processing tasks presented via computer. The exercises automatically adjust to user performance to maintain an 85% correct rate. The program will include 4 hours per week over a 10-week period for a total of up to 40 hours. The study team has support from the original developer and Posit Science. For the purposes of this trial, any participants who do not complete the total of up to 40 hours will not be counted as deviations.
  Interventions: Behavioral: Sweep Seeker; Behavioral: Bird Safari; Behavioral: Jewel Diver; Behavioral: Master Gardener; Behavioral: Road Tour
- Attention Control (Placebo Comparator): Control participants will be asked to complete activities on the computer. The program offers a choice of activities that will consist of crossword puzzles and word jumbles. The program offers a pre-determined set of computerized crossword puzzles. The site has over 100,000 puzzles and can be accessed easily via the web and are free to users. The computerized crossword puzzles do not provide for progressive challenges of increasing speed, visual field size, number of distractors or degree of difficulty of targeted stimulus differentiation. Training: Participants will be instructed to perform this active attention control intervention 4 hours per week over 10 weeks for a total of up to 40 hours, the same as BrainHQ.
  Interventions: Behavioral: Computerized Crossword Puzzles

INTERVENTIONS:
Behavioral: Sweep Seeker — The person is asked to clear the rows of blocks presented on the screen, either by moving them into horizontal or vertical blocks that have identical color. The goal is to refine and increase the response of primary visual cortex neurons and to enable the person to increase speed and accuracy of visual processing (executive function) and visual memory.
  Arms: Cognitive Training
Behavioral: Bird Safari — The user is first presented with a target bird. Subsequently, a group of birds is presented in the peripheral vision and then disappears when the trial begins. The user selects the section of the screen where the target bird appeared. The presentation speed adapts with user performance (i.e. better performance = faster presentation). The goal is to improve speed and accuracy of object identification in peripheral vision and improve visual precision important for improving memory.
  Arms: Cognitive Training
Behavioral: Jewel Diver — The person is first presented objects (jewels) on the screen. The objects are then covered with occluders (bubbles) and then identical distracters are presented. The objects move around in screen and when the movement stops, the user chooses the occluders that cover the jewels. The number of jewels adapts to performance (more jewels = better performance). The goal is to improve divided visual attention, sustained visual attention, visual working memory, and visual precision.
  Arms: Cognitive Training
Behavioral: Master Gardener — The person is presented a series of target stimuli and distracters which are presented at one time and then disappear. The locations of the stimuli are marked by icons, and the user chooses the icons where the target stimuli were once located. The goal is to increase speed and accuracy as well as the ability to extract information accurately.
  Arms: Cognitive Training
Behavioral: Road Tour — The person is presented with a target vehicle briefly in both the center of the screen and in one of eight locations in the periphery. Two vehicles are then presented briefly in the center of the screen, one of which is the target vehicle. The user must identify the location of the target vehicle in the periphery as well as identify which was the target vehicle that appeared in the center. The goal of this activity is to improve divided attention and ability to extract information and discard irrelevant information from peripheral vision.
  Arms: Cognitive Training
Behavioral: Computerized Crossword Puzzles — The program offers a pre-determined set of computerized crossword puzzles. The site has over 100,000 puzzles and can be accessed easily via the web and are free to users. The computerized crossword puzzles do not provide for progressive challenges of increasing speed, visual field size, number of distractors or degree of difficulty of targeted stimulus differentiation.
  Arms: Attention Control

SUMMARY:
For millions of cancer survivors, cognitive impairment is a prevalent, severe, and persistent problem that is associated with other symptoms (depressive symptoms, anxiety and fatigue), poorer work ability, and poorer quality of life. Available evidence, including work by the investigators own group, suggests that cognitive training may be a viable treatment option. However, to date, these studies are limited as none have been conducted in the home and therefore fail to address the transferability of these empirically based cognitive training programs to general practice.

The purpose of this translational research is to conduct a home based single-blind, randomized controlled trial to test the feasibility, satisfaction, and preliminary efficacy of cognitive training compared to attention control in breast cancer survivors (BCS) as well as to explore potential biomarkers of intervention effects.

This research innovatively builds on investigator's previous research by: 1) translating findings from the laboratory to the home setting and importantly seeks to identify facilitators and barriers of intervention use; 2) addresses limitations of previous trials (uses an attention control rather than a no-contact or wait-list control), (3) examines cognitive training effects on real-life outcomes such as associated symptoms, perceived work ability and quality of life; and (4) will be the first study in cancer survivors to explore levels of BDNF as a potentially sensitive outcome measure of intervention effects over time compared to attention control. Findings from this study will provide necessary information about the feasibility, satisfaction and preliminary efficacy of the home-based cognitive training on memory performance and processing speed as well as its effects on associated outcomes in BCS. Positive results will lead to a larger, full-scale study to determine efficacy and build evidence-based treatment for clinicians to use in treating BCS with cognitive impairment.

DETAILED DESCRIPTION:
The goal of this translational research study is to determine the feasibility, satisfaction and preliminary efficacy of cognitive training delivered in the home for cancer survivors suffering from cancer- and cancer-treatment-related cognitive impairment. In addition, this will be the first study in cancer to explore levels of brain derived neurotrophic factor (BDNF), which is now known to be associated with neural plasticity, as a potentially sensitive outcome measure of intervention effects over time compared to attention control.

Cancer- and cancer-treatment-related cognitive impairment is a national research priority. Up to 75% of the 2.6 million breast cancer survivors (BCS) living in the United States report problems with memory or feelings of mental slowness. Deficits in memory and processing speed have also been documented on neuropsychological exam and functional magnetic resonance imaging (fMRI). Cognitive impairment is a prevalent, severe, and persistent problem that is associated with other symptoms (depressive symptoms, anxiety symptoms, fatigue), poorer work ability and poorer quality of life. Cognitive training may be a viable treatment option. To date, a total of 8 pilot studies, including the investigator's own randomized controlled trial36 have noted positive effects of cognitive training in cancer survivors. These findings, combined with evidence from studies in the well elderly, suggest that cognitive training interventions to promote neuroplasticity are likely to be beneficial; however, these studies are limited as most have been conducted in the home and therefore, fail to address the transferability of these cognitive training programs to general practice. Therefore, the purpose of this translational research is to conduct a home based single-blind, randomized controlled trial to test the feasibility, satisfaction, and preliminary efficacy of cognitive training delivered in the home setting compared to attention control in breast cancer survivors (BCS). In addition, this will be the first study in cancer to explore levels of brain derived neurotrophic factor (BDNF).

Specific aims are to: (1) examine the feasibility, acceptability (facilitators and barriers) and satisfaction of the computer-based cognitive training program; (2) test the preliminary efficacy of cognitive training on improving perceived cognitive function (FACT-PCI) over time compared to attention control; (3) test the preliminary efficacy of cognitive training on improving cognitive performance (memory, processing speed, attention, working memory, executive function) over time compared to attention control; Exploratory - (1) evaluate cognitive training effects on associated outcomes (work ability, health perception status and change and quality of life) compared to attention control; and (2) explore the effect of computerized cognitive training on serum brain derived neurotrophic factor (BDNF) over time compared to attention control. BDNF is widely distributed in the brain, plays a crucial role in neuroplasticity and has been observed to correlate with cognitive function in cancer patients. A total of 68 eligible BCS will be randomized to computerized cognitive training or attention control. A blinded and trained tester will perform data collection and neuropsychological testing at two time points: baseline prior to intervention (T1) and immediately after the 10-week cognitive training -program (within 90 days) (T2). Feasibility and satisfaction will be assessed through objective indicators (study adherence, completion rate) and self-report (facilitators, barriers, and perceived satisfaction) and cognitive performance will be assessed through objective neuropsychological tests of memory, processing speed, attention, working memory, executive function assessed over the phone. In addition, the study will measure the effects of cognitive training on self-report measures of perceived cognitive function, associated symptoms (depressive symptoms, anxiety and fatigue), perceived work ability, and quality of life. Data will be analyzed using descriptive statistics and a general linear mixed model (GLMM). Simple main effects analyses will be used to follow up statistically significant interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. ≥ 21 years old at the time of informed consent
3. Ability to provide written informed consent and HIPAA authorization
4. First diagnosis of non-metastatic breast cancer.
5. Self-reported cognitive impairment
6. Subjects seeking treatment though not currently being treated or with prior treatment history for cognitive impairment.
7. ≥ 1 year post-treatment including surgery, radiation, and/or chemotherapy
8. Ability to understand, speak, read, and write English

Exclusion Criteria:

1. Comorbidities that would sufficiently impair performance or inhibit cognitive training such as: history of stroke, encephalitis, traumatic brain injury, brain surgery, dementia, or Alzheimers disease.
2. Cranial radiation or intrathecal therapy.
3. Current active major depression or substance abuse or history of bipolar disorder psychosis, schizophrenia, or learning disability.
4. History of current or other cancer except for basal cell skin cancer.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Von Ah, PhD, Principal Investigator — Ohio State University College of Nursing.; Tina Opoku, BS, Study Director — Ohio State University College of Nursing
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No identified data will be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Training: As tested in the investigator's pilot, the Brain HQ program is designed to enhance specific areas of cognitive functioning that will be tested. The goals of the Brain HQ program are to improve visual processing speed, learning and memory and attention. The exercises include time-order judgment, discrimination, spatial-match, forward-span, instruction-following, and narrative-memory tasks. This program systematically reduces the stimulus duration during a series of increasingly difficult information-processing tasks presented via computer. The exercises automatically adjust to user performance to maintain an 85% correct rate. The program will include 4 hours per week over a 10-week period for a total of up to 40 hours. The study team has support from the original developer and Posit Science. For the purposes of this trial, any participants who do not complete the total of up to 40 hours will not be counted as deviations.
  Sweep Seeker: The goal is to enable the person to increase speed and accuracy of visual processing (executive function) and visual memory.
  Bird Safari: The goal is to improve speed and accuracy of object identification in peripheral vision and improve visual precision important for improving memory.
  Jewel Diver: The goal is to improve divided visual attention, sustained visual attention, visual working memory, and visual precision.
  Master Gardener: The goal is to increase speed and accuracy as well as the ability to extract information accurately.
Period: Overall Study
Arm/Group | Cognitive Training | Attention Control
Started | 22 | 24
Completed | 19 | 17
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 1 | 5
Not completed — Illness | 2 | 2

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Attention Control | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Customized [Mean (Standard Deviation); unit: years]
  Current Age | 56.3 (9.3) | 58.8 (6.7) | 57.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 36
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 7 | 7 | 14
  White | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 19 | 17 | 36
Marital Status [Count of Participants; unit: Participants]
  Single/divorced/widowed | 8 | 4 | 12
  Married/partnered | 11 | 13 | 24
Stage of Breast Cancer [Count of Participants; unit: Participants] — Oncologists who provided the medical treatment of research participants determined the cancer stage using physical exams, clinical imaging (i.e., mammograms, ultrasounds, MRI, CT scans, PET scans, Bone Scans), clinical and pathological biopsy results, DNA testing, tumor grading and hormone receptor status tests. Higher grades of cancer were considered more advanced disease processes.
  Participants
    Stage I | 5 | 4 | 9
    Stage II | 9 | 10 | 19
    Stage III | 4 | 2 | 6
    Unsure | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire
Description: Likert-based 8-item questionnaire rating overall satisfaction, quality of training, etc. 4-point scale (range from 8-32) with higher scores indicating greater acceptability and satisfaction.
Time Frame: Within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 29.7 (6.0) | 27.9 (5.7)

2. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Abilities Between Baseline and 1 Week Post-intervention
Description: Perceived Cognitive Impairment (PCI) measured using 8-item, 5-point Likert scales with range from 8-40. The Cognitive Abilities Scale items target positive self-assessments of cognitive functioning with higher scores indicating better cognitive ability. The Cognitive Concerns Scale items are worded negatively and express concerns in the same area with higher scores indicating more cognitive concerns. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 27.9 (5.7) | 28.1 (5.4)

3. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Cognitive Concerns Between Baseline and 1 Week Post-intervention
Description: as for outcome 2
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 19.9 (6.7) | 19.9 (6.3)

4. Secondary Outcome: Change in Work Ability Index (WAI) Between Baseline and 1 Week Post-intervention
Description: Work ability was assessed by one item from the WAI. This item assessed current work ability on a Likert scale from 1 (cannot work at all) to 10 (work ability at its best) with higher scores indicating better work ability. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 7.8 (1.9) | 7.2 (2.5)

5. Secondary Outcome: Change in Medical Outcomes Study-Short-Form Health Survey (MOS SF-36) General Perceptions of Health Between Baseline and 1 Week Post-intervention
Description: General Health Perception and Quality of life (general mental health) was measured using The MOS-SF-36 with the general perceptions of health status subscale used to measure general health perceptions (5 items), on a 5-point Likert scale (total range of 5-25), with higher scores indicating positive perceptions of general health and general mental health. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 18.2 (4.6) | 18.9 (4.1)

6. Secondary Outcome: Change in Medical Outcomes Study-Short-Form Health Survey (MOS SF-36) Perceived Change in Health Between Baseline and 1 Week Post-intervention
Description: General Health Perception and Quality of life (general mental health) was measured using The MOS-SF-36 with the, changes in general health perception (1-item), on a 5-point Likert scale (total range of 1-5), with higher scores indicating positive perceptions of general health and general mental health. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 2.4 (0.9) | 2.2 (1.0)

7. Secondary Outcome: Change in Medical Outcomes Study-Short-Form Health Survey (MOS SF-36) General Mental Health Between Baseline and 1 Week Post-intervention
Description: General Health Perception and Quality of life (general mental health) was measured using The MOS-SF-36 with the general mental health (5-items), on a 5-point Likert scale (total range of 5-25), with higher scores indicating positive perceptions of general health and general mental health. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 5.3 (1.0) | 5.4 (1.2)

8. Other Pre Specified Outcome: Change in Rey Auditory Verbal Learning Test (Rey AVLT) Total Between Baseline and 1 Week Post-intervention
Description: Measure of learning and episodic memory. List of 15 words given and asked to recall, score range from 0-75. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 53.8 (6.8) | 56.7 (8.2)

9. Other Pre Specified Outcome: Change in Rey Auditory Verbal Learning Test (Rey AVLT) Delayed Between Baseline and 1 Week Post-intervention
Description: Measure of delayed memory. List of 15 words given and asked to recall at delayed timeframe, score range from 0-15. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 9.8 (2.8) | 12.3 (2.4)

10. Other Pre Specified Outcome: Change in Rivermead Behavioral Paragraph Recall Test Between Baseline and 1 Week Post-intervention
Description: Measure of immediate memory. 14-item test with score range from 0-12. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 7.4 (3.3) | 8.3 (3.2)

11. Other Pre Specified Outcome: Change in Rivermead Behavioral Paragraph Recall Test -Delayed Between Baseline and 1 Week Post-intervention
Description: Measure of delayed memory. 14-item test with score range from 0-12. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 6.7 (3.3) | 7.9 (3.1)

12. Other Pre Specified Outcome: Change in Symbol Digit Modalities Test [SDMT], Oral Response Version Between Baseline and 1 Week Post-intervention
Description: Measure of speed of processing. 90 seconds to pair numbers and figures, score range 0-110. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 53.6 (9.3) | 58.1 (7.4)

13. Other Pre Specified Outcome: Change in Digit Span, Total Raw Score From the WAIS-III Between Baseline and 1 Week Post-intervention
Description: Measures attention and working memory by asking participants to Repeat a number sequence, The total score being calculated by adding the correct responses from both the "Digits Forward" and "Digits Backward" sections, with each correct sequence contributing one point. Scores range from 0 to 32. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 17.3 (3.0) | 17.7 (3.7)

14. Other Pre Specified Outcome: Change in Controlled Oral Word Association (COWA) Between Baseline and 1 Week Post-intervention
Description: Measure of verbal/executive functioning. Provide a spontaneous list of words within 60 seconds, score range from 0-60. Higher scores indicate better outcomes. Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
score on a scale | 43.0 (9.8) | 46.4 (9.3)

15. Other Pre Specified Outcome: Change in Serum Levels of Brain-Derived Neurotropic Factor (BDNF) Between Baseline and 1 Week Post-intervention
Description: Plasma levels of BDNF were measured in duplicate by ELISA (catalog number DBD00; R&D Systems, Minneapolis, MN). The minimum detectable level of BDNF in this assay is 20 pg/ ml, and the within-assay variation is 4.2% at 1339 pg/ml. Higher levels indicate higher concentrations of BDNF (reported in pg/ml). Outcomes are controlled for the baseline assessment.
Time Frame: Baseline and within 1 week post-intervention
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Cognitive Training | Attention Control
Number analyzed (Participants) | 19 | 17
pg/ml | 22,404 (7287.8) | 24,920 (6277.4)

ADVERSE EVENTS:
Time Frame: 10 Week period of study intervention
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Cognitive Training | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05570604/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT05570604/ICF_001.pdf